CLINICAL TRIAL: NCT03075891
Title: Efficacy Comparison of Ivermectin 1% Topical Cream Associated With Doxycycline 40 mg Modified Release (MR) Capsules Versus Ivermectin 1% Topical Cream Associated With Placebo in the Treatment of Severe Rosacea
Brief Title: Oracea Soolantra Association in Participants With Severe Rosacea
Acronym: ANSWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.113322
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2019-11-29 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2019-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin; Doxycycline; Capsules

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivermectin 1% cream + Doxycycline 40 mg MR capsules (Experimental)
  Interventions: Drug: Ivermectin 1% cream; Drug: Doxycycline 40 mg MR (30 mg Immediate Release & 10 mg Delayed Release beads) capsules
- Ivermectin 1% cream + Oral placebo capsules (Placebo Comparator)
  Interventions: Drug: Ivermectin 1% cream; Other: Oral placebo capsules

INTERVENTIONS:
Drug: Ivermectin 1% cream — Topical to the face, approximately one small pea size amount per facial region (right and left cheeks, forehead, chin, and nose) once a day for 12 weeks
Drug: Doxycycline 40 mg MR (30 mg Immediate Release & 10 mg Delayed Release beads) capsules — 1 Capsule once-daily for 12 weeks
  Arms: Ivermectin 1% cream + Doxycycline 40 mg MR capsules
Other: Oral placebo capsules — 1 Capsule once-daily for 12 weeks
  Arms: Ivermectin 1% cream + Oral placebo capsules

SUMMARY:
The main objective of this study is to evaluate the efficacy of Ivermectin 1% topical cream associated with Doxycycline 40 mg Modified release (MR) capsules versus Ivermectin 1% topical cream associated with Placebo in the treatment of severe Rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject age ≥ 18 years or older;
* Subject with a minimum of 20 but not more than 70 inflammatory lesions (papules and pustules) of rosacea on the face at Baseline visit;
* Subject with severe rosacea with papulopustular lesions (according to the Investigator's Global Assessment (IGA) score rated 4);
* Female subjects of childbearing potential with a negative urine pregnancy test (UPT);
* Female subjects of childbearing potential must practice a highly effective method of contraception during the study.

Exclusion Criteria:

* Subjects with particular forms of rosacea or other concomitant facial dermatoses that may be confounded with rosacea;
* Subjects with more than 2 nodules of rosacea on the face;
* Subjects with any uncontrolled chronic or serious disease or medical condition that may either interfere with the interpretation of the clinical trial results, or with optimal participation in the study or would present a significant risk to the subject;
* Subjects with known or suspected allergies or sensitivities to any component of the investigational and non-investigational products, including the active ingredients doxycycline and ivermectin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (8):
  - Private Practice, Fort Smith, Arkansas
  - Private practice, Sacramento, California
  - Private practice, Boca Raton, Florida
  - Private practice, Louisville, Kentucky
  - Private Practice, Metairie, Louisiana
  - Private practice, Omaha, Nebraska
  - Private practice, Las Vegas, Nevada
  - Private practice, Pflugerville, Texas
- Canada (5):
  - Private practice, Markham
  - Private practice, Montreal
  - Private practice, Peterborough
  - Private practice, Richmond Hill
  - Private practice, Waterloo
- Hungary (7):
  - Private practice, Budapest
  - University, Debrecen
  - Hospital, Miskolc
  - Private practice, Pécel
  - University, Pécs
  - University, Szeged
  - Private practice, Szolnok

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 sites in Canada, Czech Republic, Germany, Hungary, Poland, and United States of America between 05 July 2017 to 08 February 2018.
Pre-assignment Details: A total of 273 participants were randomized and treated, out of which 251 participants completed the study.
Groups:
- Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules: Ivermectin 1% (percent) cream: Topical to the face, approximately one small pea size amount per facial region (right and left cheeks, forehead, chin, and nose) once a day for 12 weeks.
  Doxycycline 40 mg (milligram) Modified Release (MR) (30 mg Immediate Release & 10 mg Delayed Release beads) capsules: 1 Capsule once-daily for 12 weeks.
Period: Overall Study
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Started | 135 | 138
Completed | 126 | 125
Not Completed | 9 | 13
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 3 | 1
Not completed — visits not performed (no time) | 1 | 0
Not completed — Drug abuse relapse issue | 0 | 1
Not completed — Participant requiring study withdrawal | 0 | 1
Not completed — Adverse event, non-fatal | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of the entire population enrolled and randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules | Total
Number analyzed (Participants) | 135 | 138 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 110 | 219
  >=65 years | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.5) | 51.6 (13.3) | 52 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 80 | 155
  Male | 60 | 58 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 133 | 136 | 269
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Skin phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to VI. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly; skin phototype IV = light brown skin, burns minimally, always tans well; skin phototype V = brown skin, rarely burns, tans profusely; skin phototype VI = dark brown or black skin, never burns, tans profusely.
  Participants
    Skin phototype I | 5 | 11 | 16
    Skin phototype II | 82 | 83 | 165
    Skin phototype III | 37 | 38 | 75
    Skin phototype IV | 8 | 6 | 14
    Skin phototype V | 1 | 0 | 1
    Skin phototype VI | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Inflammatory Lesion Count at Week 12
Description: Percent change from baseline in inflammatory lesion count at week 12 was reported. Inflammatory lesions included facial inflammatory lesions of rosacea (that is [i.e.] papules and pustules) which were defined as follows: Papule - a small, solid elevation less than 1.0 centimeter (cm) in diameter; and Pustule - a small, circumscribed elevation of the skin, which contains yellow white exudates. Papules and pustules were counted separately on each of the 5 facial regions (forehead, chin, nose, right cheek and left cheek). Notably, nodules (i.e. circumscribed, elevated, solid lesions more than 1.0 cm in diameter with palpable depth) were not included in the count of inflammatory lesions.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) population consisted of the entire population enrolled and randomized. The last observation carried forward (LOCF) method was used to impute missing values for inflammatory lesion count.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percent change | -80.29 (21.65) | -73.56 (30.52)
Statistical Analysis 1: Comparison: Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules vs Ivermectin 1% Cream + Oral Placebo Capsules; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count at Weeks 4 and 8
Description: Percent change from baseline in inflammatory lesion count at Weeks 4 and 8 was reported. Inflammatory lesions included facial inflammatory lesions of rosacea (i.e. papules and pustules) which were defined as follows: Papule - a small, solid elevation less than 1.0 centimeter in diameter. Pustule - a small, circumscribed elevation of the skin, which contains yellow white exudates. Papules and pustules were counted separately on each of the 5 facial regions (forehead, chin, nose, right cheek and left cheek). Notably, nodules (i.e. circumscribed, elevated, solid lesions more than 1.0 cm in diameter with palpable depth) were not included in the count of inflammatory lesions.
Time Frame: Baseline, Weeks 4 and 8
Population: ITT population consisted of the entire population enrolled and randomized. The LOCF method was used to impute missing values for inflammatory lesion count.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percent change
  Week 4 | -48.15 (26.71) | -39.27 (27.93)
  Week 8 | -69.14 (24.10) | -61.44 (28.74)

3. Secondary Outcome: Percentage of Participants With Clear Inflammatory Lesions at Week 12
Description: Percentage of participants with clear inflammatory lesions at week 12 was reported. Inflammatory lesions included facial inflammatory lesions of rosacea (i.e. papules and pustules) which were defined as follows: Papule - a small, solid elevation less than 1.0 cm in diameter. Pustule - a small, circumscribed elevation of the skin, which contains yellow white exudates. Papules and pustules were counted separately on each of the 5 facial regions (forehead, chin, nose, right cheek and left cheek). Notably, nodules (i.e. circumscribed, elevated, solid lesions more than 1.0 cm in diameter with palpable depth) were not included in the count of inflammatory lesions.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants | 17.8 | 7.2

4. Secondary Outcome: Percentage of Participants With 100 Percent (%) Reduction in Inflammatory Lesions at Weeks 4, 8 and 12
Description: Percentage of participants with 100% reduction in inflammatory lesions at Weeks 4, 8 and 12 was reported. Inflammatory lesions included facial inflammatory lesions of rosacea (i.e. papules and pustules) which were defined as follows: Papule - a small, solid elevation less than 1.0 centimeter in diameter. Pustule - a small, circumscribed elevation of the skin, which contains yellow white exudates. Papules and pustules were counted separately on each of the 5 facial regions (forehead, chin, nose, right cheek and left cheek). Notably, nodules (i.e. circumscribed, elevated, solid lesions more than 1.0 cm in diameter with palpable depth) were not included in the count of inflammatory lesions.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Week 4: Yes | 1.5 | 0.0
  Week 4: No | 98.5 | 100.0
  Week 8: Yes | 5.2 | 2.9
  Week 8: No | 94.8 | 97.1
  Week 12: Yes | 17.8 | 7.2
  Week 12: No | 82.2 | 92.8

5. Secondary Outcome: Clinician's Erythema Assessment (CEA) Total Score at Weeks 4, 8 and 12
Description: The evaluator assessed the participant's diffuse persistent facial erythema of rosacea by performing a static ("snap shot") evaluation of erythema severity at a social distance of approximately 50 centimeter (cm) using CEA scale, at each visit. CEA is a 5 point scale where 0 = clear (clear skin with no signs of erythema); 1 = almost clear (almost clear; slight redness); 2 = mild (mild erythema; definite redness); 3 = moderate (moderate erythema; marked redness); 4 = severe (severe erythema; fiery redness). A higher score than baseline indicates a worse outcome.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
Units on a scale
  Week 4 | 2.47 (0.94) | 2.56 (0.94)
  Week 8 | 1.85 (0.95) | 1.97 (0.94)
  Week 12 | 1.51 (1.02) | 1.58 (0.95)

6. Secondary Outcome: Percentage of Participants in Each Clinician's Erythema Assessment Score Category at Weeks 4, 8 and 12
Description: as for outcome 5
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Week 4 (0= Clear skin) | 0.7 | 0.7
  Week 4 (1= Almost clear) | 16.3 | 12.3
  Week 4 (2= Mild erythema) | 31.9 | 34.1
  Week 4 (3= Moderate erythema) | 37.8 | 36.2
  Week 4 (4= Severe erythema) | 13.3 | 16.7
  Week 8 (0= Clear skin) | 5.2 | 1.4
  Week 8 (1= Almost clear) | 31.1 | 33.3
  Week 8 (2= Mild erythema) | 43.7 | 39.1
  Week 8 (3= Moderate erythema) | 13.3 | 18.8
  Week 8 (4= Severe erythema) | 6.7 | 7.2
  Week 12 (0= Clear skin) | 14.1 | 7.2
  Week 12 (1= Almost clear) | 41.5 | 47.8
  Week 12 (2= Mild erythema) | 28.1 | 29.7
  Week 12 (3= Moderate erythema) | 11.9 | 10.1
  Week 12 (4= Severe erythema) | 4.4 | 5.1

7. Secondary Outcome: Investigator's Global Assessment (IGA) Total Score at Weeks 4, 8 and 12
Description: The evaluator assessed the participant's rosacea by performing a static ("snap shot") evaluation, at a social distance of approximately 50 cm, using the IGA score. IGA is a 5 point scale where, 0 = clear (no inflammatory lesions present, no erythema); 1 = almost clear (very small papules/pustules, very mild erythema present); 2 = mild (few small papules/pustules, mild erythema); 3 = moderate (severe small or large papules/pustules, moderate erythema); 4 = severe (numerous small and/or large papules/pustules, severe erythema).
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
Units on a scale
  Week 4 | 2.59 (0.88) | 2.84 (0.83)
  Week 8 | 1.78 (0.83) | 2.04 (0.93)
  Week 12 | 1.34 (0.89) | 1.57 (0.95)

8. Secondary Outcome: Percentage of Participants in Each Investigator's Global Assessment Score Category at Weeks 4, 8 and 12
Description: as for outcome 7
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Week 4 (0 - Clear) | 1.5 | 0.7
  Week 4 (1 - Almost clear) | 11.1 | 5.1
  Week 4 (2- Mild) | 25.2 | 23.9
  Week 4 (3 - Moderate) | 51.9 | 50.0
  Week 4 (4 - Severe) | 10.4 | 20.3
  Week 8 (0 - Clear) | 3.0 | 3.6
  Week 8 (1 - Almost clear) | 34.8 | 22.5
  Week 8 (2 - Mild) | 48.1 | 47.8
  Week 8 (3 - Moderate) | 9.6 | 18.1
  Week 8 (4 - Severe) | 4.4 | 8.0
  Week 12 (0 - Clear) | 11.9 | 5.1
  Week 12 (1 - Almost clear) | 54.8 | 54.3
  Week 12 (2 - Mild) | 24.4 | 26.1
  Week 12 (3 - Moderate) | 5.2 | 8.0
  Week 12 (4 - Severe) | 3.7 | 6.5

9. Secondary Outcome: Stinging/Burning Severity Score at Weeks 4, 8 and 12
Description: The evaluator recorded the severity of the participant's facial stinging/burning sensation during the last 24 hours according to the stinging/burning scale. Stinging/burning scale is a 4 point scale where, 0 = none (No stinging/burning ); 1 = mild (slight warm, tingling/stinging sensation, not really bothersome); 2 = moderate (definite warm, tingling/stinging sensation that is somewhat bothersome); 3 = severe (hot, tingling/stinging sensation that has caused definite discomfort).
Time Frame: Weeks 4, 8 and 12
Population: ITT population consisted of the entire population enrolled and randomized. The LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
units on a scale
  Week 4 | 0.73 (0.79) | 0.65 (0.75)
  Week 8 | 0.41 (0.64) | 0.44 (0.67)
  Week 12 | 0.31 (0.55) | 0.33 (0.63)

10. Secondary Outcome: Percentage of Participants in Each Stinging/Burning Severity Score Category at Weeks 4, 8 and 12
Description: as for outcome 9
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Week 4 (0 - None) | 47.4 | 50.0
  Week 4 (1 - Mild) | 32.6 | 36.2
  Week 4 (2 - Moderate) | 19.3 | 12.3
  Week 4 (3 - Severe) | 0.7 | 1.4
  Week 8 (0 - None) | 67.4 | 64.5
  Week 8 (1 - Mild) | 24.4 | 28.3
  Week 8 (2 - Moderate) | 8.1 | 5.8
  Week 8 (3 - Severe) | 0.0 | 1.4
  Week 12 (0 - None) | 73.3 | 75.4
  Week 12 (1 - Mild) | 22.2 | 17.4
  Week 12 (2 - Moderate) | 4.4 | 6.5
  Week 12 (3 - Severe) | 0.0 | 0.0

11. Secondary Outcome: Global Improvement Total Score at Week 12 (Last Visit/Early Termination)
Description: Participants were evaluated for his/her improvement in rosacea compared to his/her rosacea condition before study, using global Improvement scale. It is a 7 item scale where, 0=complete improvement (all signs and symptoms of disease have resolved [100% improvement]); 1=excellent improvement (nearly all signs and symptoms cleared [90% improvement]. Only minimal residual signs and symptoms remain); 2=very good improvement (majority of the signs and symptoms have resolved [about 75% improvement]); 3=good improvement (significant improvement, but many signs and symptoms remain [about 50% improvement]); 4=minimal improvement (slight overall improvement, but not clinically significant [about 25% improvement]); 5=no change (overall severity similar to baseline); 6=worse (worse than baseline).
Time Frame: Week 12 (last visit/early termination)
Population: ITT population consisted of the entire population enrolled and randomized. Here the over all number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 126 | 129
units on a scale | 1.79 (1.20) | 1.81 (1.20)

12. Secondary Outcome: Percentage of Participants in Each Global Improvement Score Category at Week 12 (Last Visit/Early Termination)
Description: Participants were to evaluated for his/her improvement in rosacea compared to his/her rosacea condition before study, using global Improvement scale. it is a 7 item scale where, 0=complete improvement (all signs and symptoms of disease have resolved [100% improvement]); 1=excellent improvement (nearly all signs and symptoms cleared [90% improvement]. Only minimal residual signs and symptoms remain); 2=very good improvement (majority of the signs and symptoms have resolved [about 75% improvement]); 3=good improvement (significant improvement, but many signs and symptoms remain [about 50% improvement]); 4=minimal improvement (slight overall improvement, but not clinically significant [about 25% improvement]); 5=no change (overall severity similar to baseline); 6=worse (worse than baseline). .
Time Frame: Week 12 (last visit/early termination)
Population: ITT population consisted of the entire population enrolled and randomized. Here the overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 126 | 129
percentage of participants
  0 - Complete improvement | 7.9 | 6.2
  1 - Excellent improvement | 39.7 | 44.2
  2 - Very good improvement | 31.7 | 25.6
  3 - Good improvement | 11.9 | 15.5
  4 - Minimal improvement | 4.0 | 3.9
  5 - No change | 4.0 | 3.9
  6 - Worse | 0.8 | 0.8

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily had a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE was any untoward medical occurrence that at any dose: results in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: From the signing of the informed consent form (ICF) up to Week 12
Population: Safety population (all participants treated [APT]) - consisted of the ITT population, after exclusion of participants who never used the treatment with certainty based on monitoring report.
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
Participants
  Adverse Events | 27 | 50
  Serious Adverse Events | 1 | 1

14. Secondary Outcome: Dermatology Life Quality Index (DLQI) Questionnaire Total Score at Week 12 (Last Visit/Early Termination Visit)
Description: DLQI focuses on impact of dermatological diseases on quality of life. It is a 10-item validated quality-of-life questionnaire specific to dermatological conditions. 1) how itchy, sore, painful, stinging?, 2) how embarrassed/self-conscious?, 3) interfere shopping or looking after home or garden?, 4) Influence clothes?, 5) affect social/leisure activity?, 6) difficult to do sport?, 7) prevent from working/studying? or If no, problem at work/studying?, 8) problem with partner or close friend?, 9) cause sexual difficulties?, 10) problem caused by treatment?. Total score ranged from 0-30 (each question had a score range of 0- 3) where, 0-1=no effect at all on life; 2-5=small effect on life; 6-10=moderate effect on life; 11- 20=very large effect on life; 21-30=extremely large effect on life. A higher score indicates a low quality of life due to more severe disease.
Time Frame: Week 12 (last visit/early termination)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 125 | 129
units on a scale | 1.4 (2.2) | 2.2 (4.0)

15. Secondary Outcome: Percentage of Participants in Each Dermatology Life Quality Index (DLQI) Questionnaire Score Category
Description: Impact of study treatments on subjects' quality of life was measured by using DLQI questionnaire. DLQI focuses on impact of dermatological diseases on quality of life. It is a 10-item validated quality-of-life questionnaire specific to dermatological conditions. 1) how itchy, sore, painful, stinging?, 2) how embarrassed/self-conscious?, 3) interfere shopping or looking after home or garden?, 4) Influence clothes?, 5) affect social/leisure activity?, 6) difficult to do sport?, 7) prevent from working/studying? or If no, problem at work/studying?, 8) problem with partner or close friend?, 9) cause sexual difficulties?, 10) problem caused by treatment?. Total score ranged from 0-30 (each question had a score range of 0- 3) where, 0-1=no effect at all on life; 2-5=small effect on life; 6-10=moderate effect on life; 11- 20=very large effect on life; 21-30=extremely large effect on life. A higher score indicates a low quality of life due to more severe disease.
Time Frame: Baseline, Week 12 (last visit/early termination)
Population: ITT population consisted of the entire population enrolled and randomized. Here, n, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Baseline: 0-1 | 17.8 | 18.8
  Baseline: 2-5 | 37.8 | 33.3
  Baseline: 6-10 | 27.4 | 32.6
  Baseline: 11-20 | 14.8 | 12.3
  Baseline: 21-30 | 2.2 | 2.9
  Week 12: 0-1 | 68.0 | 65.1
  Week 12: 2-5: number analyzed (Participants) | 125 | 129
  Week 12: 2-5 | 26.4 | 24.0
  Week 12: 6-10: number analyzed (Participants) | 125 | 129
  Week 12: 6-10 | 4.8 | 7.0
  Week 12: 11-20: number analyzed (Participants) | 125 | 129
  Week 12: 11-20 | 0.8 | 3.1
  Week 12: 21-30: number analyzed (Participants) | 125 | 129
  Week 12: 21-30 | 0.0 | 0.8

16. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index Questionnaire Total Score at Week 12 (Last Visit/Early Termination)
Description: Percent Change from Baseline in Dermatology Life Quality Index questionnaire Total Score at Last Visit. DLQI focuses on impact of dermatological diseases on quality of life. It is a 10-item validated quality-of life questionnaire specific to dermatological conditions. 1) how itchy, sore, painful, stinging?, 2) how embarrassed/self-conscious?, 3) interfere shopping or looking after home or garden?, 4) Influence clothes?, 5) affect social/leisure activity?, 6) difficult to do sport?, 7) prevent from working/studying? or If no, problem at work/studying?, 8) problem with partner or close friend?, 9) cause sexual difficulties?, 10) problem caused by treatment?. Total score ranged from 0-30 (each question had a score range of 0-3) where, 0-1=no effect at all on life; 2-5=small effect on life; 6-10=moderate effect on life; 11- 20=very large effect on life; 21-30=extremely large effect on life. A higher score indicates a low quality of life due to more severe disease.
Time Frame: Baseline, Week 12 (last visit/early termination)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 120 | 126
Percent Change | -59.5 (66.3) | -59.2 (70.6)

17. Secondary Outcome: EuroQol-5 Dimension-5 Level (EQ-5D-5L) Questionnaire at Week 12 (Last Visit/Early Termination Visit)
Description: EQ-5D-5L is a 5-level, 5-dimensional format standardized instrument for use as a measure of health outcome used to assess the impact of study treatments on participants quality of life as follows: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression. Each dimension comprised of 5 levels with corresponding numeric scores, where 1 indicated no problems, and 5 indicated extreme problems. Participant selected answer for each of 5 dimensions considering response that best matches his/her health today with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). An increase in the EQ-5D-5L total score indicates improvement.
Time Frame: Week 12/Last visit or early termination visit
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 125 | 129
units on a scale | 83.5 (16.2) | 83.0 (15.1)

18. Secondary Outcome: Percentage of Participants in Each EuroQol-5 Dimension-5 Level Questionnaire Questions Who Reported No Problems at Baseline and Week 12 (Last Visit/Early Termination)
Description: as for outcome 17
Time Frame: Baseline, Week 12 (last visit/early termination)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 135 | 138
percentage of participants
  Baseline: Mobility | 80 | 84.1
  Baseline: Self-care | 96.3 | 97.8
  Baseline: Usual activities | 85.9 | 89.1
  Baseline: Pain/discomfort | 55.6 | 57.2
  Baseline: Anxiety/depression | 65.9 | 69.6
  Week 12: Mobility: number analyzed (Participants) | 125 | 129
  Week 12: Mobility | 80.0 | 83.7
  Week 12: Self-care: number analyzed (Participants) | 125 | 129
  Week 12: Self-care | 94.4 | 96.9
  Week 12: Usual activities: number analyzed (Participants) | 125 | 129
  Week 12: Usual activities | 89.6 | 90.7
  Week 12: Pain/discomfort: number analyzed (Participants) | 125 | 129
  Week 12: Pain/discomfort | 68.0 | 79.1
  Week 12: Anxiety/depression: number analyzed (Participants) | 125 | 129
  Week 12: Anxiety/depression | 77.6 | 82.2

19. Secondary Outcome: Percentage of Participants Reported Work Productivity and Activity Impairment: General Health (WPAI:GH) Questionnaire for Currently Employed Question at Week 12 (Last Visit/Early Termination Visit)
Description: WPAI:GH questionnaire was an instrument to measure impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Low scores indicate little or no impact of health problems on work and activities, and a negative change in the WPAI score indicates improvement. Currently Employed question was assessed in this outcome measure.
Time Frame: Week 12 (Last visit/early termination visit)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 125 | 128
percentage of participants
  No | 34.1 | 34.8
  Yes | 65.9 | 65.2

20. Secondary Outcome: Work Productivity and Activity Impairment: General Health (WPAI:GH) Questionnaire - Hours Missed at Work, Impact to Productivity at Work and Daily Activities at Week 12
Description: WPAI:GH questionnaire is an instrument to measure impairment in both paid and unpaid work during the past week including questions: missed hours from work because of rosacea?, missed hours from work because of other reason?, number of Working hours. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Low scores indicate little or no impact of health problems on work and activities, and a negative change in the WPAI score indicates improvement.
Time Frame: Week 12 (Last visit/Early termination visit)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 80 | 82
hours
  Missed hours from work because of rosacea | 0.1 (0.9) | 0.0 (0.0)
  Missed hours from work because of other reason | 4.2 (10.9) | 2.9 (9.6)
  Number of Working hours | 36.3 (17.7) | 38.2 (14.8)

21. Secondary Outcome: Work Productivity and Activity Impairment: General Health (WPAI:GH) Questionnaire (How Much Rosacea Affect Productivity at Work, How Much Rosacea Affect Daily Activity) at Week 12 (Last Visit/Early Termination Visit)
Description: WPAI:GH questionnaire is an instrument to measure impairment in both paid and unpaid work during the past week, on a scale ranging from 0 (health problems had no effect) to 10 (health problems completely prevented them from working) including questions: 5) how much rosacea affect productivity at work?; 6) how much rosacea affect daily activity?. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Low scores indicated little or no impact of health problems on work and activities, and a negative change in the WPAI score indicated improvement."
Time Frame: Week 12 (Last visit/Early termination visit)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 125 | 128
units on a scale
  How much rosacea affect productivity at work | 0.6 (1.5) | 0.5 (1.2)
  How much rosacea affect daily activity | 0.5 (1.3) | 0.7 (1.5)

22. Secondary Outcome: Percentage of Participants Who Reported Satisfied for Subject Satisfaction Questionnaire at Week 12 (Last Visit/Early Termination Visit): Part A
Description: Subject's satisfaction questionnaire was used to specifically collect the subjects' feedback on the treatment regimen, the level of satisfaction and future usage. Questionnaire consisted of 4 parts: Part A, B, C and D. where Part A consisted of following 12 questions about study drugs (capsules and cream): 1-Time the study regimen took to work, 2-Improvement of facial lesions, 3-Improvement of facial redness, 4-Improvement of ocular symptoms, 5-Improvement of flushing episodes, 6-How bothered by side effects, 7-Your face looks, 8-You feel, 9-Easy to incorporate in daily routine, 10-Using the study regimen again, 11-Overall satisfaction, 12-Compared to last treatment. Satisfied score of questionnaire meant as participants responded as Very satisfied (Questions-1,2,3,4,5,11), Not bothered at all (Question-6), A lot better (Questions- 7,8,12), yes (Question-10), strongly agree (Question-9).
Time Frame: Week 12 (Last visit/early termination visit)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 125 | 129
percentage of participants
  1.Time the study regimen took to work | 48.0 | 45.0
  2.Improvement of facial lesions | 48.0 | 46.5
  3.Improvement of facial redness | 45.6 | 41.1
  4.Improvement of ocular symptoms | 25.6 | 26.4
  5.Improvement of flushing episodes | 41.6 | 38.0
  6.How bothered by side effects | 84.0 | 76.7
  7.Your face looks | 70.4 | 65.9
  8.You feel | 61.6 | 55.0
  9.Easy to incorporate in daily routine | 62.4 | 58.9
  10.Using the study regimen again | 86.4 | 82.9
  11.Overall satisfaction | 54.4 | 52.7
  12.Compared to last treatment | 42.4 | 41.1

23. Secondary Outcome: Percentage of Participants Who Reported Strongly Agree for Subject Satisfaction Questionnaire at Week 12 (Last Visit/Early Termination Visit): Part B
Description: Part B of Questionnaire consisted of following 10 questions about both provided skin care products cleanser and moisturizer: 1-Easy to incorporate into a daily routine, 2-Recommend to my family or friends, 3-Help my skin look healthier, 4-More confident with rosacea, 5-More confident with skin appearance, 6-Positive difference in the appearance, 7-Keep using both skin care products, 8-Make my skin more hydrated, 9-Improve the texture of my skin, 10-Pleasant to use.
Time Frame: Week 12 (Last visit/early termination visit)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 124 | 129
percentage of participants
  1.Easy to incorporate into a daily routine | 68.5 | 70.5
  2.Recommend to my family or friends | 60.5 | 52.7
  3.Help my skin look healthier | 58.1 | 50.4
  4.More confident with rosacea | 33.1 | 32.6
  5.More confident with skin appearance | 37.9 | 36.4
  6.Positive difference in the appearance | 47.6 | 44.2
  7.Keep using both skin care products | 52.4 | 48.8
  8.Make my skin more hydrated | 42.7 | 38.8
  9.Improve the texture of my skin | 35.5 | 34.9
  10.Pleasant to use | 54.0 | 50.4

24. Secondary Outcome: Percentage of Participants Who Reported Strongly Agree for Subject Satisfaction Questionnaire at Week 12 (Last Visit/Early Termination Visit): Part C
Description: Part C subject satisfaction questionnaire consisted of following 4 questions about the cosmetic product cleanser: 1-Clean healthy skin feeling, 2-Deep cleansing without stripping moisture, 3-Rinsed off easily, 4-Not make my skin feel tight or dry.
Time Frame: Week 12 (Last visit or early termination visit)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 124 | 129
percentage of participants
  1.Clean healthy skin feeling | 49.2 | 46.5
  2.Deep cleansing without stripping moisture | 41.1 | 40.3
  3.Rinsed off easily | 54.0 | 48.8
  4.Not make my skin feel tight or dry | 59.7 | 50.4

25. Secondary Outcome: Percentage of Participants Who Reported Strongly Agree for Subject Satisfaction Questionnaire at Week 12 (Last Visit/Early Termination Visit): Part D
Description: Part D of subject satisfaction questionnaire consisted of following 4 questions about the cosmetic product moisturizer: 1-Skin feel soft and smooth, 2-Improve my skin moisture, 3-Leave my skin hydrated and protected, 4-Provide comforting sensation.
Time Frame: Week 12 (Last visit/early termination visit)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
Number analyzed (Participants) | 123 | 129
percentage of participants
  1.Skin feel soft and smooth | 48.0 | 35.7
  2.Improve my skin moisture | 38.2 | 34.1
  3.Leave my skin hydrated and protected | 42.3 | 38.0
  4.Provide comforting sensation | 43.9 | 37.2

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form (ICF) up to week 12
Description: Safety population (all participants treated [APT]) - consisted of the ITT population, after exclusion of participants who never used the treatment with certainty based on monitoring report.
Arm/Group | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules | Ivermectin 1% Cream + Oral Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/138
Serious Adverse Events (participants affected / at risk) | 1/135 | 1/138
Other Adverse Events (participants affected / at risk) | 17/135 | 33/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules (N=135) | Ivermectin 1% Cream + Oral Placebo Capsules (N=138)
Multilevel discopathy in the cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholezystolithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin 1% Cream + Doxycycline 40 mg MR Capsules (N=135) | Ivermectin 1% Cream + Oral Placebo Capsules (N=138)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol: Version for all countries except Germany (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03075891/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT03075891/SAP_001.pdf